CLINICAL TRIAL: NCT05297240
Title: Retrospective Study of the Use of Belantamab Mafodotin (Blenrep®) in Patients With Relapsed and/or Refractory Multiple Myeloma (RRMM) in Spain.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: PETHEMA Foundation (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: GEM-RELAMAB
Record Dates: First submitted 2022-03-17; First posted 2022-03-28 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: RELAPSED AND/OR REFRACTORY MULTIPLE MYELOMA
MeSH Terms: interventions — belantamab mafodotin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Belantamab mafodotin — At least one dose of belantamab mafodotin as part of the compassionate use or the expanded access program in Spain between November 2019 and June 2021.

SUMMARY:
The proposal of this study is to retrospectively analyze the experience with belantamab mafodotin monotherapy in patients with RRMM included in the compassionate use or in the expanded access program in Spain between November 2019 and June 2021.

The focus of the study will be on the estimation of the magnitude of the treatment effect as assessed by the overall response rate (ORR), duration of response (DOR), progression free survival (PFS), overall survival (OS), and the safety of single agent belantamab mafodotin in patients with RRMM.

Subjects may receive treatment until progression. Myeloma disease status will be evaluated locally for response and progression per International Myeloma Working Group (IMWG) criteria from cycle 1 day 1 until confirmed progressive disease, death, unacceptable toxicity, or lost to follow-up (whichever occurs first).

DETAILED DESCRIPTION:
The proposal of this study is to retrospectively analyze the experience with belantamab mafodotin monotherapy in patients with RRMM included in the compassionate use or in the expanded access program in Spain between November 2019 and June 2021.

Subjects may receive treatment until progression. Myeloma disease status will be evaluated locally for response and progression per International Myeloma Working Group (IMWG) criteria from cycle 1 day 1 until confirmed progressive disease, death, unacceptable toxicity, or lost to follow-up (whichever occurs first).

The study has the following objectives:

Primary objective

- The primary objective of this study is to evaluate the efficacy of belantamab mafodotin in terms of overall response, and the different response categories when administered as a single agent in patients with RRMM.

Secondary objectives:

* Describe the safety and tolerability of single-agent belantamab mafodotin.
* The overall incidence of ophthalmologic complications.
* Estimate duration of response (DOR).
* Estimate time to response (TTR).
* Estimate time to next treatment (TTNT).
* Estimate progression-free survival (PFS) and overall survival (OS).
* Type of treatment administered after single-agent belantamab mafodotin and estimate PFS2.

ELIGIBILITY:
Inclusion Criteria:

* Reception of at least one dose of belantamab mafodotin as part of the compassionate use or the expanded access program in Spain between November 2019 and June 2021

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Every patient receiving at least one dose of belantamab mafodotin as part of the compassionate use or the expanded access program in Spain between November 2019 and June 2021 will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2022-03-24 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | Throughout the study period. Approximately 3 years
  The percentage of participants with the best overall confirmed response: partial response (PR), very good partial response (VGPR), complete response (CR), or stringent complete response (sCR).
  per International Myeloma Working Group (IMWG) uniform response criteria.

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events (AEs) | Throughout the study period. Approximately 3 years
  Number and percentage of treatment-emergent adverse events (AEs)
Incidence of ocular events | Throughout the study period. Approximately 3 years
  Number and percentage of ocular events
Duration of response (DOR) | Throughout the study period. Approximately 3 years
  The time from first date of PR or better to date of disease progression or death due to any cause.
Time to response (TTR) | Throughout the study period. Approximately 3 years
  The time from date of first dose of belantamab mafodotin to date of first occurrence of response.
Time to next treatment (TTNT). | Throughout the study period. Approximately 3 years
  The time from first dose of belantamab mafodotin to first day when subject receives another myeloma treatment.
Progression free survival (PFS) | Throughout the study period. Approximately 3 years
  The time from start of treatment until progression or death from any cause
Overall survival (OS) | Throughout the study period. Approximately 3 years
  The time from start of treatment until death from any cause.
Second progression free survival (PFS2) | Throughout the study period. Approximately 3 years
  The time from start of belantamab mafodotin to progression on next-line treatment, or death from any cause, whichever is earlier; otherwise censored at the last time known to be alive and without second objective disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Javier de la Rubia, Principal Investigator — Hospital La Fe de Valencia; Adrián Alegre, Principal Investigator — Hospital La Princesa (Madrid); María Victoria Mateos, Principal Investigator — Hospital Clínico, Salamanca
Locations (62):
- Spain (62):
  - H. Universitario de Albacete, Albacete
  - H. Doctor José Molina Orosa, Arrecife
  - H. San Agustín, Avilés
  - H. Ntra. Señora Sonsoles, Ávila
  - H. Clinic de Barcelona, Barcelona
  - H. Moises Broggi, Barcelona
  - H. Vall d' Hebron, Barcelona
  - H. Basurto, Bilbao
  - H. Cruces, Bilbao
  - H. Calahorra, Calahorra
  - H. Reina Sofía, Córdoba
  - H. General Elche, Elche
  - H. Fuenlabrada, Fuenlabrada
  - H. Galdakao, Galdakao
  - H. Francisco de Borja, Gandia
  - ICO Girona, Girona
  - H. Un. Virgen de las Nieves, Granada
  - H. Un. Guadalajara, Guadalajara
  - H. Juan Ramón Jiménez, Huelva
  - H. Universitario de Jaén, Jaén
  - H. Un. Doctor Negrín, Las Palmas de Gran Canaria
  - H. Severo Ochoa, Leganés
  - H. León, León
  - H. San Pedro, Logroño
  - H. Un. Lucus Augusti, Lugo
  - Fundación Jiménez Díaz, Madrid
  - H. Gregorio Marañón, Madrid
  - H. Moncloa, Madrid
  - H. Ruber Juan Bravo, Madrid
  - H. Un. Doce de Octubre, Madrid
  - H. Un. Infanta Sofía, Madrid
  - H. Un. La Paz, Madrid
  - H. Un. La Princesa, Madrid
  - H. Un. Puerta del Hierro, Madrid
  - H. Un. Quirón Salud, Madrid
  - H.M. Sanchinarro, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario Henares, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - H. Virgen de la Victoria, Málaga
  - H. Rey Juan Carlos, Móstoles
  - H. Morales Meseguer, Murcia
  - H. Un. Virgen de la Arrixaca, Murcia
  - H. Universitario Central Asturias, Oviedo
  - H. Son Llatzer, Palma de Mallorca
  - H. Un. Son Espases, Palma de Mallorca
  - H. Montecelo, Pontevedra
  - H. Un. Salamanca, Salamanca
  - H. Un. Canarias, Santa Cruz de Tenerife
  - H. Un. Marqués de Valdecilla, Santander
  - H. General Segovia, Segovia
  - H. Un. Virgen de Valme, Seville
  - H. Virgen del Rocío, Seville
  - H. Mutua Terrasa, Terrassa
  - H. Ntra. Señora del Prado, Toledo
  - H. Un. Torrejón, Torrejón de Ardoz
  - H. Un. Dr. Peset, Valencia
  - H. Universitario de la Fe, Valencia
  - H. Universitario de Valladolid, Valladolid
  - H. Clinico Un. Lozano Blesa, Zaragoza
  - H. Miguel Servet, Zaragoza
  - H. Royo Villanova, Zaragoza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Palumbo A, Anderson K. Multiple myeloma. N Engl J Med. 2011 Mar 17;364(11):1046-60. doi: 10.1056/NEJMra1011442. No abstract available. PMID 21410373
- [Background] Kumar SK, Dispenzieri A, Lacy MQ, Gertz MA, Buadi FK, Pandey S, Kapoor P, Dingli D, Hayman SR, Leung N, Lust J, McCurdy A, Russell SJ, Zeldenrust SR, Kyle RA, Rajkumar SV. Continued improvement in survival in multiple myeloma: changes in early mortality and outcomes in older patients. Leukemia. 2014 May;28(5):1122-8. doi: 10.1038/leu.2013.313. Epub 2013 Oct 25. PMID 24157580
- [Background] Zanwar S, Abeykoon JP, Kapoor P. Challenges and Strategies in the Management of Multiple Myeloma in the Elderly Population. Curr Hematol Malig Rep. 2019 Apr;14(2):70-82. doi: 10.1007/s11899-019-00500-4. PMID 30820879
- [Background] Kumar SK, Callander NS, Hillengass J, Liedtke M, Baljevic M, Campagnaro E, Castillo JJ, Chandler JC, Cornell RF, Costello C, Efebera Y, Faiman M, Garfall A, Godby K, Holmberg L, Htut M, Huff CA, Kang Y, Landgren O, Malek E, Martin T, Omel J, Raje N, Sborov D, Singhal S, Stockerl-Goldstein K, Tan C, Weber D, Johnson-Chilla A, Keller J, Kumar R. NCCN Guidelines Insights: Multiple Myeloma, Version 1.2020. J Natl Compr Canc Netw. 2019 Oct 1;17(10):1154-1165. doi: 10.6004/jnccn.2019.0049. PMID 31590151
- [Background] Hoyos V, Borrello I. The immunotherapy era of myeloma: monoclonal antibodies, vaccines, and adoptive T-cell therapies. Blood. 2016 Sep 29;128(13):1679-87. doi: 10.1182/blood-2016-05-636357. Epub 2016 Aug 9. PMID 27506540
- [Background] Rickert RC, Jellusova J, Miletic AV. Signaling by the tumor necrosis factor receptor superfamily in B-cell biology and disease. Immunol Rev. 2011 Nov;244(1):115-33. doi: 10.1111/j.1600-065X.2011.01067.x. PMID 22017435
- [Background] Frigyesi I, Adolfsson J, Ali M, Christophersen MK, Johnsson E, Turesson I, Gullberg U, Hansson M, Nilsson B. Robust isolation of malignant plasma cells in multiple myeloma. Blood. 2014 Feb 27;123(9):1336-40. doi: 10.1182/blood-2013-09-529800. Epub 2014 Jan 2. PMID 24385542
- [Background] Tai YT, Mayes PA, Acharya C, Zhong MY, Cea M, Cagnetta A, Craigen J, Yates J, Gliddon L, Fieles W, Hoang B, Tunstead J, Christie AL, Kung AL, Richardson P, Munshi NC, Anderson KC. Novel anti-B-cell maturation antigen antibody-drug conjugate (GSK2857916) selectively induces killing of multiple myeloma. Blood. 2014 May 15;123(20):3128-38. doi: 10.1182/blood-2013-10-535088. Epub 2014 Feb 25. PMID 24569262
- [Background] Seckinger A, Delgado JA, Moser S, Moreno L, Neuber B, Grab A, Lipp S, Merino J, Prosper F, Emde M, Delon C, Latzko M, Gianotti R, Luoend R, Murr R, Hosse RJ, Harnisch LJ, Bacac M, Fauti T, Klein C, Zabaleta A, Hillengass J, Cavalcanti-Adam EA, Ho AD, Hundemer M, San Miguel JF, Strein K, Umana P, Hose D, Paiva B, Vu MD. Target Expression, Generation, Preclinical Activity, and Pharmacokinetics of the BCMA-T Cell Bispecific Antibody EM801 for Multiple Myeloma Treatment. Cancer Cell. 2017 Mar 13;31(3):396-410. doi: 10.1016/j.ccell.2017.02.002. Epub 2017 Mar 2. PMID 28262554
- [Background] Moreaux J, Legouffe E, Jourdan E, Quittet P, Reme T, Lugagne C, Moine P, Rossi JF, Klein B, Tarte K. BAFF and APRIL protect myeloma cells from apoptosis induced by interleukin 6 deprivation and dexamethasone. Blood. 2004 Apr 15;103(8):3148-57. doi: 10.1182/blood-2003-06-1984. Epub 2003 Dec 4. PMID 15070697
- [Background] Tai YT, Acharya C, An G, Moschetta M, Zhong MY, Feng X, Cea M, Cagnetta A, Wen K, van Eenennaam H, van Elsas A, Qiu L, Richardson P, Munshi N, Anderson KC. APRIL and BCMA promote human multiple myeloma growth and immunosuppression in the bone marrow microenvironment. Blood. 2016 Jun 23;127(25):3225-36. doi: 10.1182/blood-2016-01-691162. Epub 2016 Apr 28. PMID 27127303
- [Background] Sanchez E, Li M, Kitto A, Li J, Wang CS, Kirk DT, Yellin O, Nichols CM, Dreyer MP, Ahles CP, Robinson A, Madden E, Waterman GN, Swift RA, Bonavida B, Boccia R, Vescio RA, Crowley J, Chen H, Berenson JR. Serum B-cell maturation antigen is elevated in multiple myeloma and correlates with disease status and survival. Br J Haematol. 2012 Sep;158(6):727-38. doi: 10.1111/j.1365-2141.2012.09241.x. Epub 2012 Jul 18. PMID 22804669
- [Background] Lee L, Bounds D, Paterson J, Herledan G, Sully K, Seestaller-Wehr LM, Fieles WE, Tunstead J, McCahon L, Germaschewski FM, Mayes PA, Craigen JL, Rodriguez-Justo M, Yong KL. Evaluation of B cell maturation antigen as a target for antibody drug conjugate mediated cytotoxicity in multiple myeloma. Br J Haematol. 2016 Sep;174(6):911-22. doi: 10.1111/bjh.14145. Epub 2016 Jun 17. PMID 27313079
- [Background] Trudel S, Lendvai N, Popat R, Voorhees PM, Reeves B, Libby EN, Richardson PG, Anderson LD Jr, Sutherland HJ, Yong K, Hoos A, Gorczyca MM, Lahiri S, He Z, Austin DJ, Opalinska JB, Cohen AD. Targeting B-cell maturation antigen with GSK2857916 antibody-drug conjugate in relapsed or refractory multiple myeloma (BMA117159): a dose escalation and expansion phase 1 trial. Lancet Oncol. 2018 Dec;19(12):1641-1653. doi: 10.1016/S1470-2045(18)30576-X. Epub 2018 Nov 12. PMID 30442502
- [Background] Lonial S, Lee HC, Badros A, Trudel S, Nooka AK, Chari A, Abdallah AO, Callander N, Lendvai N, Sborov D, Suvannasankha A, Weisel K, Karlin L, Libby E, Arnulf B, Facon T, Hulin C, Kortum KM, Rodriguez-Otero P, Usmani SZ, Hari P, Baz R, Quach H, Moreau P, Voorhees PM, Gupta I, Hoos A, Zhi E, Baron J, Piontek T, Lewis E, Jewell RC, Dettman EJ, Popat R, Esposti SD, Opalinska J, Richardson P, Cohen AD. Belantamab mafodotin for relapsed or refractory multiple myeloma (DREAMM-2): a two-arm, randomised, open-label, phase 2 study. Lancet Oncol. 2020 Feb;21(2):207-221. doi: 10.1016/S1470-2045(19)30788-0. Epub 2019 Dec 16. PMID 31859245
- [Background] Lonial S, Lee HC, Badros A, et al. Cancer. 2021 Jul 27. doi: 10.1002/cncr.33809. Online ahead of print. PMID: 34314018
- [Background] Shah JJ, Abonour R, Gasparetto C, Hardin JW, Toomey K, Narang M, Srinivasan S, Kitali A, Zafar F, Flick ED, Rifkin RM. Analysis of Common Eligibility Criteria of Randomized Controlled Trials in Newly Diagnosed Multiple Myeloma Patients and Extrapolating Outcomes. Clin Lymphoma Myeloma Leuk. 2017 Sep;17(9):575-583.e2. doi: 10.1016/j.clml.2017.06.013. Epub 2017 Jun 17. PMID 28886839
- [Background] Chari A, Romanus D, Palumbo A, Blazer M, Farrelly E, Raju A, Huang H, Richardson P. Randomized Clinical Trial Representativeness and Outcomes in Real-World Patients: Comparison of 6 Hallmark Randomized Clinical Trials of Relapsed/Refractory Multiple Myeloma. Clin Lymphoma Myeloma Leuk. 2020 Jan;20(1):8-17.e16. doi: 10.1016/j.clml.2019.09.625. Epub 2019 Oct 10. PMID 31722839
- [Background] Fiala M, et al. The real-world characteristics and outcomes of newly diagnosed myeloma patients ineligible for clinical trials. Clin. Lymphoma Myeloma Leuk. 2017;17:e55-e56
- [Background] Hungria VTM, et al. Real-world (RW) multiple myeloma (MM) patients (Pts) remain under-represented in clinical trials based on standard laboratory parameters and baseline characteristics: analysis of over 3,000 Pts from the Insight MM Global, Prospective, Observational Study. Blood. 2019;134:1887a
- [Background] Klausen TW, Gregersen H, Abildgaard N, Andersen NF, Frolund UC, Gimsing P, Helleberg C, Vangsted AJ. The majority of newly diagnosed myeloma patients do not fulfill the inclusion criteria in clinical phase III trials. Leukemia. 2019 Feb;33(2):546-549. doi: 10.1038/s41375-018-0272-0. Epub 2018 Sep 28. No abstract available. PMID 30267010
- [Background] Bergin K, McQuilten Z, Moore E, Wood E, Spencer A. Myeloma in the Real World: What Is Really Happening? Clin Lymphoma Myeloma Leuk. 2017 Mar;17(3):133-144.e1. doi: 10.1016/j.clml.2016.12.002. Epub 2016 Dec 26. PMID 28153487
- [Background] Song X, Cong Z, Wilson K. Real-world treatment patterns, comorbidities, and disease-related complications in patients with multiple myeloma in the United States. Curr Med Res Opin. 2016;32(1):95-103. doi: 10.1185/03007995.2015.1105202. Epub 2015 Nov 20. PMID 26488820
- [Background] Kumar S, Paiva B, Anderson KC, Durie B, Landgren O, Moreau P, Munshi N, Lonial S, Blade J, Mateos MV, Dimopoulos M, Kastritis E, Boccadoro M, Orlowski R, Goldschmidt H, Spencer A, Hou J, Chng WJ, Usmani SZ, Zamagni E, Shimizu K, Jagannath S, Johnsen HE, Terpos E, Reiman A, Kyle RA, Sonneveld P, Richardson PG, McCarthy P, Ludwig H, Chen W, Cavo M, Harousseau JL, Lentzsch S, Hillengass J, Palumbo A, Orfao A, Rajkumar SV, Miguel JS, Avet-Loiseau H. International Myeloma Working Group consensus criteria for response and minimal residual disease assessment in multiple myeloma. Lancet Oncol. 2016 Aug;17(8):e328-e346. doi: 10.1016/S1470-2045(16)30206-6. PMID 27511158